CLINICAL TRIAL: NCT00949494
Title: Pilot Trial of Effects of Intra-articular Synvisc Therapy on Cartilage Determined by dGEMRIC in Patients With OA of the Knee
Brief Title: Effects of Synvisc on Cartilage in Knee Osteoarthritis (OA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); Northwestern University (Other)
Responsible Party: Principal Investigator, Pottumarthi Prasad, Associate Director Department of Radiology Center for Advanced MR Research, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: EH 06-159
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis
Keywords: knee osteoarthritis, synvisc, hyaluronan, dGEMRIC,cartilage
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synvisc (Active Comparator)
  Interventions: Device: Synvisc
- Placebo (Placebo Comparator)
  Interventions: Device: Synvisc

INTERVENTIONS:
Device: Synvisc — intra-articular, 3 weekly injections
  Other Names: hyaluronan

SUMMARY:
Hylan G-F 20 (Synvisc) is an FDA-approved hyaluronate derivative used to treat knee osteoarthritis (OA). Animal studies have shown that Synvisc can have favorable effects on cartilage when injected into joints. This study attempts to evaluate the effects of Synvisc when injected into knees of patients with knee OA by means of a specialized MRI technology (dGEMRIC).

DETAILED DESCRIPTION:
Hylan G-F 20 (Synvisc) is an FDA-approved hyaluronate derivative which is administered by injection into osteoarthritic joints for the treatment of osteoarthritis. Preclinical investigations have demonstrated that Hylan G-F 20 can favorably affect chondrocyte metabolism and recent clinical studies [Ann Rheum Dis. 2004 May;63(5):478-82; Osteoarthritis Cartilage. 2005 Mar;13(3):216-24] provide support for a disease-modifying effect of Hylan G-F 20 therapy. This study will utilize dGEMRIC imaging of patients with knee OA to assess the effects of Hylan G-F 20 therapy on cartilage in vivo over time. Delayed Gadolinium Enhanced MRI of the Cartilage (dGEMRIC) permits a quantitative assessment of GAG distribution within intact cartilage in vivo. Since dGEMRIC is noninvasive, the technique may be useful to non-invasively monitor the influence of various treatments on hyaline cartilage.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 40 to 80 years of age who meet the ACR Criteria for osteoarthritis of the knee.
2. Radiographic evidence of OA, Kellgren and Lawrence grade I to III on prior X-rays (taken within 6 months of the screening visit) or at screening. Only the tibio-femoral joint will be evaluated (patello-femoral disease will not be considered).
3. Mild to moderate levels of knee pain as determined by a VAS pain score of 3-6/10 that has been stable for at least 1 month prior to screening visit.
4. Stable management regimen for knee OA pain for at least 1 month prior to screening visit. Subjects can be managed by physical measures alone, simple analgesics, NSAIDs, nutriceuticals or other agents with no significant change in treatment regimen during the 1 month prior to screening visit.
5. Ability to comply with the requirements of the study
6. Able to maintain stable exercise/activity program during course of the study

6. Signed and dated consent form 7. Women of child-bearing potential should agree to the use of an appropriate method of contraception and have a confirmed negative pregnancy test at screening.

Exclusion Criteria:

1. Radiographic evidence of Kellgren and Lawrence grade IV OA
2. Knee pain <3 or >6 out of 10 on VAS pain scale.
3. Change in management regimen for knee OA during the preceding month.
4. Subjects with any metal implant such as cardiac pacemakers, spinal cord stimulators or bionic ear devices.
5. Subjects who are unable to receive gadolinium contrast agent injection because of contraindications.
6. Unable to undergo an MRI exam because of contraindication, e.g. claustrophobia.
7. Inflammatory arthritis, e.g. rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus.
8. History of other diseases that may involve the study joint including inflammatory joint disease, crystalline disease, endocrinopathies, metabolic disease, knee infection of the chosen knee, neuropathic disorders, avascular necrosis, Paget's disease or tumors
9. Recent trauma to study joint.
10. Known loose bodies in the study joint.
11. Patients taking oral steroids.
12. Patients with active malignancy.
13. Patients who are either high-performance athletes or, in the opinion of the investigator, are highly sedentary and not likely to ambulate at least 20-30 minutes/day.
14. In the opinion of the investigator, the subject has an unstable medical condition.
15. Participating in another study or has participated in a study evaluating investigational drugs, devices or biologics within three months of enrollment in this study.
16. Study subject has ever previously received hyaluronan therapy.
17. Arthroscopic or open surgery to the study joint within the previous twelve months.
18. Anticipated need for knee surgery to the study joint.
19. History of joint replacement, intra-articular fracture, osteotomy, arthroplasty or meniscectomy of the study knee.
20. Intra-articular injection of corticosteroid to study joint within the past six months.
21. Morbid obesity defined as BMI of greater than 40.
22. Study subject has known sensitivity to any component of Hylan G-F 20 including bird feathers, eggs or poultry.
23. Subject has an active systemic infection.
24. Subject on coumadin or other anticoagulant.
25. Musculoskeletal pain that may preclude the subject from remaining motionless for the MRI exam.
26. Women who are pregnant or lactating.
27. Subjects with "clinically significant" malalignment.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Percent change in dGEMRIC Index (T1(Gd)) in femoral and tibial compartments | 3 and 6 months

SECONDARY OUTCOMES:
Subjects' global assessment of disease using a 10 point Likert scale | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pottumarthi V Prasad, PhD, Principal Investigator — Endeavor Health
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Northshore University Hospital, Evanston, Illinois